CLINICAL TRIAL: NCT01020448
Title: Prostate Cancer Antigen-3 (PCA-3) and TMPRSS2-ERG (T2-ERG) Score Changes During Initiation of Androgen Deprivation Therapy (ADT) With Triptorelin 22.5mg in Patients With Advanced Prostate Cancer (PCA): A Phase III, Single Arm Multicentre Study
Brief Title: Effect of Triptorelin (Decapeptyl®) 22.5 mg on Two Biomarkers in Patients With Advanced Prostate Cancer
Acronym: Triptocare
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8-79-52014-168; 2009-012786-58 (EudraCT Number)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Results first posted 2015-07-15 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: Locally advanced or metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triptorelin (Decapeptyl®) 22.5 mg (Experimental)
  Interventions: Drug: Triptorelin (Decapeptyl®)

INTERVENTIONS:
Drug: Triptorelin (Decapeptyl®) — One intramuscular injection of triptorelin (Decapeptyl®) 22.5mg performed once all baseline procedures and assessments have been completed.

SUMMARY:
The purpose of this study is to evaluate the effect of an initial hormonal treatment gonadotrophin-releasing hormone (GnRH Agonist) on 2 biomarkers (PCA3 and TMPRSS2-ERG), in patients with histologically confirmed and advanced stages of prostate cancer. Their characteristics, according to risk factors such as PSA and Gleason score will be determined at baseline and 1, 3 and 6 month post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* A histologically confirmed, locally advanced or metastatic prostate cancer, and naïve to androgen deprivation therapy, and a candidate for hormonal treatment.
* An estimated survival time of at least twelve months according to the investigator's assessment.
* A performance status score ≤ 2 according to the World Health Organisation (WHO) criteria.

Exclusion Criteria:

* Previous surgical castration.
* Previous or has planned curative prostate cancer therapy (radiation/surgery)
* Previous hormone therapy (GnRH analogues, estrogens or anti-androgens)
* Patients with risk of a serious complication in the case of tumour flare (vertebral metastases threatening spinal cord compression or significant obstructive uropathy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (59):
- Belgium (6):
  - Hôpital Erasme, Brussels
  - UZ Brussels, Brussels
  - UCL Saint-Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
- Denmark (4):
  - Fredericia Sygehus, Fredericia
  - Frederiksbergs Hospital, Frederiksberg
  - Herlev University Hospital, Herlev
  - Odense Universitets hospital, Odense
- France (15):
  - Clinique Rhône Durance, Avignon
  - Hôpital Pellegrin, Bordeaux
  - CHU Henri Mondor, Créteil
  - CHU Michalon, Grenoble
  - Chru Lille, Lille
  - Hôpital Nord, Marseille
  - Clinique Beau Soleil, Montpellier
  - Private practice, Nancy
  - CHU Nantes, Nantes
  - CHU Pasteur, Nice
  - Hôpital Val de Grâce, Paris
  - Institut Mutualiste Monsouris, Paris
  - Hôpital Henry Gabrielle, Saint-Genis-Laval
  - Hôpital Foch, Suresnes
  - CHU Toulouse, Toulouse
- Italy (2):
  - IRCCS Fondazione S. Raffaele del Monte Tabor, Milan
  - AOU San Luigi Gonzaga, Torino
- Latvia (2):
  - P.Stradins Clinical University Hospital, Riga
  - Center of Oncology, Riga
- Lithuania (3):
  - Medical University Clinics, Kaunas
  - University Hospital, Klaipėda
  - University Oncological Institute, Vilnius
- Netherlands (4):
  - Ziekenhuis Amstelland, Amstelveen
  - Academisch Medisch Centrum, Amsterdam
  - Diaconessenhuis, Leiden
  - Antonius Ziekenhuis, Sneek
- Romania (4):
  - Medical Center, Arad
  - Oncology Institute, Bucharest
  - Sc E-Uro Srl, Cluj-Napoca
  - Oncomed, Timișoara
- Spain (8):
  - Hospital Juan Canalejo, A Coruña
  - Hospital Valle Hebrón, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital General Universitario, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Infanta Sofía, Madrid
  - Instituto de Oncología, Valencia
- United Kingdom (11):
  - Bristol Royal Infirmary, Bristol
  - Addenbrookes Hospital, Cambridge
  - University Hospital Wales, Cardiff
  - University Hospital Coventry, Coventry
  - Derby City Hosptial, Derby
  - Royal Devon and Exeter Hospital, Exeter
  - Falkirk & District Royal Infirmary, Falkirk
  - Leicester General Hospital, Leicester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Lister Hospital, Stevenage

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date: 30-Nov-2009. Subjects screened were 339 and screen failures were 13.
Groups:
- Triptorelin (Decapeptyl®) 22.5 mg: Triptorelin (Decapeptyl®): One intramuscular injection of triptorelin (Decapeptyl®) 22.5 mg performed once all baseline procedures and assessments have been completed.
Period: Pre-assignment
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Started | 339
Completed | 326
Not Completed | 13
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 5
Not completed — Does Not Meet Entry Criteria | 2
Period: Treatment
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Started | 325 (One patient was excluded from the safety population as no post-baseline assessment was available)
Completed | 299
Not Completed | 26
Not completed — Adverse Event | 11
Not completed — Consent Withdrawn | 3
Not completed — Disease Progression | 2
Not completed — Lack of Efficacy | 8
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Number analyzed (Participants) | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 325
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 307
  More than one race | 0
  Unknown or Not Reported | 10
Height [Mean (Standard Deviation); unit: Cm] | 172.3 (6.5)
Weight [Mean (Standard Deviation); unit: KG] | 79.6 (13.4)
BMI [Mean (Standard Deviation); unit: kg/m²] | 26.79 (4.23)
PCA-3 Score [Number; unit: participants] — PCA-3 score = (mRNA PCA3/mRNA PSA)x1000
  * Non-assessable = Associated PSA mRNA <7500 copies/mL
  * ≤BLQ = PCA-3 mRNA is below the concentration of the calibrator and associated PSA mRNA >7500 copies/mL
  * <35 = PCA-3 mRNA above BLQ and less than 35
  * ≥35 = PCA-3 mRNA greater or equal to 35
  participants
    Non-assessable | 39
    ≤BLQ | 15
    <35 | 89
    ≥35 | 179
    Missing - No sample analysis done | 3

OUTCOME MEASURES:

1. Primary Outcome: PCA3 Score Expressed as a Ratio of PCA3 mRNA (Messenger Ribonucleic Acid) Over PSA (Prostate Specific Antigen) mRNA
Description: PCA-3 score = (mRNA PCA3/mRNA PSA)x1000
  * Non-assessable = Associated PSA mRNA <7500 copies/mL
  * ≤BLQ = PCA-3 mRNA is below the concentration of the calibrator and associated PSA mRNA >7500 copies/mL
  * <35 = PCA-3 mRNA above BLQ and less than 35
  * ≥35 = PCA-3 mRNA greater or equal to 35
Time Frame: At month 6 post-treatment
Population: Number of participants analyzed were 298 as one participant was admitted to an asylum and was withdrawn before month 1 visit was scheduled. No post-baseline assessment was available for this patient.
Measure: Number; unit: participants
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Number analyzed (Participants) | 298
participants
  Non-assessable | 232
  ≤BLQ | 27
  <35 | 10
  ≥35 | 24
  Missing - No sample analysis done | 5

2. Secondary Outcome: PCA3 Score Expressed as a Ratio of PCA3 mRNA Over PSA mRNA
Description: as for outcome 1
Time Frame: At month 1 and 3 post-treatment
Population: Analysis based on number (N) of patients with a valid value. Intention-to-treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Number analyzed (Participants) | 322
participants
  Month 1: Non-assessable (N=322) | 109
  Month 1: ≤BLQ (N=322) | 40
  Month 1: <35 (N=322) | 80
  Month 1: ≥35 (N=322) | 91
  Month 1: Missing - No sample analysis done (N=322) | 2
  Month 3: Non-assessable (N=313) | 215
  Month 3: ≤BLQ (N=313) | 31
  Month 3: <35 (N=313) | 34
  Month 3: ≥35 (N=313) | 31
  Month 3: Missing - No sample analysis done (N=313) | 2

3. Secondary Outcome: TMPRSS2-ERG Score (Expressed as a Ratio of T2-ERG mRNA Over PSA mRNA)
Description: TMPRSS2-ERG = (TMPRSS2-ERG mRNA / PSA mRNA) x 100000
  A TMPRSS2-ERG score <35 was described as 'negative' and a TMPRSS2-ERG score ≥35 as 'positive.'
Time Frame: At baseline, month 1, 3 and 6 post-treatment
Population: Analysis based on number (N) of patients with a valid value. ITT population.
Measure: Number; unit: participants
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Number analyzed (Participants) | 322
participants
  Baseline: Non-assessable (N=322) | 33
  Baseline: <35 negative (N=322) | 140
  Baseline: ≥35 positive (N=322) | 149
  Month 1: Non-assessable (N=322) | 117
  Month 1: <35 negative (N=322) | 97
  Month 1: ≥35 positive (N=322) | 106
  Month 1: Missing - No sample analysis done (N=322) | 2
  Month 3: Non-assessable (N=313) | 213
  Month 3: <35 negative (N=313) | 45
  Month 3: ≥35 positive (N=313) | 53
  Month 3: Missing - No sample analysis done (N=313) | 2
  Month 6: Non-assessable (N=298) | 241
  Month 6: <35 negative (N=298) | 24
  Month 6: ≥35 positive (N=298) | 27
  Month 6: Missing - No sample analysis done (N=298) | 6

4. Secondary Outcome: Proportion of Patients Medically Castrated (i.e. With Serum Testosterone Levels of <50 ng/dL)
Time Frame: At month 1, 3 and 6 post-treatment
Population: Analysis based on number (N) of patients with a valid value. ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Number analyzed (Participants) | 322
percentage of participants
  Month 1 (N=322) | 94.7
  Month 3 (N=313) | 95.2
  Month 6 (N=298) | 90.9

5. Secondary Outcome: PSA Level
Time Frame: At baseline, month 1, 3 and 6 post-treatment
Population: Analysis based on number (N) of patients with a valid value. ITT population.
Measure: Median (Full Range); unit: μg/L
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Number analyzed (Participants) | 322
μg/L
  Baseline (N=321) | 45.4 [1 to 12239]
  Month 1 (N=320) | 8.3 [0 to 581]
  Month 3 (N=311) | 1.8 [0 to 969]
  Month 6 (N=296) | 1.2 [0 to 1251]

6. Secondary Outcome: Safety, Assessed Through the Collection of Adverse Events (AEs)
Time Frame: For the duration of the study (up to month 6)
Measure: Number; unit: participants
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Number analyzed (Participants) | 325
participants
  Any Adverse Events (AEs) | 193
  Any Treatment Emergent Adverse Events (TEAEs) | 190
  TEAEs Leading to Withdrawal | 11
  TEAEs Leading to Death | 11
  Serious Adverse Events (SAEs) | 37

ADVERSE EVENTS:
Time Frame: Up to month 6
Arm/Group | Triptorelin (Decapeptyl®) 22.5 mg
Serious Adverse Events (participants affected / at risk) | 37/325
Other Adverse Events (participants affected / at risk) | 89/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triptorelin (Decapeptyl®) 22.5 mg (N=325)
Fall (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Heart failure (Cardiac disorders) | 2
Chronic heart failure (Cardiac disorders) | 1
Perforated colon (Gastrointestinal disorders) | 1
Perforated gall bladder (Gastrointestinal disorders) | 1
Fecal peritonitis (Gastrointestinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Liver failure (Hepatobiliary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Septicaemia (Infections and infestations) | 1
Suicide (Psychiatric disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Urosepsis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Worsening of chronic lumbago (Musculoskeletal and connective tissue disorders) | 1
Severe anemia (Blood and lymphatic system disorders) | 2
Paraplegia (Nervous system disorders) | 1
Cancer progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone pain due to metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectum tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fever (General disorders) | 1
Entero-cutaneous fistula (Gastrointestinal disorders) | 1
Septic venous thrombophlebitis (General disorders) | 1
Septicemia due to catheter (Infections and infestations) | 1
Urothelial tumor in the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Claudication (Vascular disorders) | 1
Asthenia (General disorders) | 1
Weight gain (Investigations) | 1
Acute pneumonia (Infections and infestations) | 2
Appendicitis acute (Infections and infestations) | 1
Urethral stricture (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Blocked nephrostomy catheter (General disorders) | 1
Sudden death (General disorders) | 1
Allergy to conc med (Immune system disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Right pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Right central pulmonary tumor malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Cardio respiratory arrest (Cardiac disorders) | 1
Larynx adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonia pneumocystis (Infections and infestations) | 1
Thoracic pain (General disorders) | 1
Unspecific thoracic pain (General disorders) | 1
Hemorrhage prostate (Reproductive system and breast disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Right inguinal hernia (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Chest infection (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Depression (Psychiatric disorders) | 1
Deliberate medication overdose (Injury, poisoning and procedural complications) | 1
End stage renal failure (Renal and urinary disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Heamaturia (Renal and urinary disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Increased pain in right thigh (Musculoskeletal and connective tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin (Decapeptyl®) 22.5 mg (N=325)
Hot flush (Vascular disorders) | 89 (89)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No